CLINICAL TRIAL: NCT00467896
Title: A Comparison of Safety and Inhalation Times of Ventavis (Iloprost) Inhalation Solution Delivered by I-Neb Utilizing Power Disc-6 and Power Disc-15 "Power 15 Study"
Brief Title: The "Power 15 Study": Safety Study of Inhalation of Ventavis With the Power Disc-15 Setting
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C200-008
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Pulmonary Hypertension
Keywords: PAH; iloprost; Ventavis; Pulmonary Arterial Hypertension; Actelion Pharmaceuticals; Cotherix
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Iloprost

ARMS (1):
- Iloprost (Experimental): The study enrolled patients who were already using iloprost (10 µg/mL) standard dose (5 µg) delivered by I-neb® Adaptive Aerosol Delivery (AAD) System with Power Disc-6 (PD-6) without any safety or tolerability concerns, thereby facilitating a direct comparison with the Power Disc-15 (PD-15). The single arm design allowed each patient to serve as his/her own control.
  Interventions: Drug: Iloprost PD-6; Drug: Iloprost PD-15

INTERVENTIONS:
Drug: Iloprost PD-6 — Period I: Patients received iloprost administered using PD-6 for the 37 days prior to the first dosing of iloprost using PD-15. Iloprost inhalation solution was delivered using the I-neb® AAD System. Patients were required to use their own I-neb®.
  Other Names: Ventavis
Drug: Iloprost PD-15 — Period II: Iloprost inhalation solution was delivered using the investigational product PD-15 with I-neb® AAD System for 37 days. Patients were required to use their own I-neb®.
  Other Names: Ventavis

SUMMARY:
A Comparison of Safety and Inhalation Times of Ventavis (iloprost) Inhalation Solution delivered by I-Neb Utilizing Power Disc-6 and Power Disc-15 "Power 15 Study"

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-85 years
* Have a current diagnosis of symptomatic pulmonary arterial hypertension (PAH) classified by one of the following: a) idiopathic pulmonary arterial hypertension (IPAH) or familial pulmonary arterial hypertension (FPAH); b) PAH associated with one of the following connective tissue diseases and mild or no lung parenchymal disease: scleroderma spectrum of disease, systemic lupus erythematosis, or mixed connective tissue disease, c) PAH associated with repaired atrial septal defect (ASD), ventricular septal defect (VSD), or patent ductus arteriosis (PDA) ≥ 1 year post-operative from Screening, d) PAH associated with human immunodeficiency virus (HIV), or e) PAH associated with the use of anorexigens (e.g. fenfluramine-phentermine)
* On a stable and well tolerated dose regimen of Ventavis (5 μg per dose) for at least 4 weeks prior to the Screening visit, using the I-neb AAD System equipped with Power Disc-6

Exclusion Criteria:

* Receipt of any prostacyclin or prostacyclin analogue other than Ventavis within the 12 weeks preceding the Screening visit
* Receipt of atrial septostomy within the 6 months preceding Screening
* History of left-sided heart disease
* Clinically relevant obstructive lung disease
* Chronic renal or liver disease
* Uncontrolled systemic hypertension or hypotension
* Cerebrovascular event within the 6 months preceding Screening

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-09; Primary Completion 2010-11 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Mathier, MD, Principal Investigator — University of Pittsburgh Medical Center; Ramagopal Tumuluri, MD, Principal Investigator — Aurora Medical Group - Cardiovascular Services; Charles J. Burch, MD, Principal Investigator — Diagnostic Research Group; David Baratz, MD, Principal Investigator — Pulmonary Associates; Ben DeBoisblanc, MD, Principal Investigator — Ochsner Health System; Adaani Frost, MD, Principal Investigator — Baylor College of Medicine; Victor Test, MD, Principal Investigator — UCSD Medical Center, Thorton Hospital; Sif Handsdottir, MD, Principal Investigator — University of Iowa Hospital & Clinics; Myung Park, MD, Principal Investigator — University of Maryland Hospital; Evelyn Horn, MD, Principal Investigator — New York Presbyterian Hospital; Erika Berman-Rosenzweig, MD, Principal Investigator — Columbia University; Victor Tapson, MD, Principal Investigator — Duke University
Locations (12):
- United States (12):
  - Pulmonary Associates, Phoenix, Arizona
  - UCSD Medical Center, Thorton Hospital, La Jolla, California
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Hospital, Baltimore, Maryland
  - Columbia University Medical Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Diagnostic Research Group, San Antonio, Texas
  - Aurora Medical Group - Cardiovascular Services, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled across 12 U.S. centers.
Pre-assignment Details: Adults with symptomatic pulmonary arterial hypertension (PAH) who were using Ventavis (Iloprost) Inhalation Solution Delivered by I-Neb Utilizing Power Disc-6 (PD-6) were enrolled
Groups:
- Iloprost: iloprost (10 µg/mL) standard dose (5 µg) delivered by I-neb® Adaptive Aerosol Delivery System (AAD) using Power Disc-6 (PD-6) and Power Disc-15 (PD-15).
Period: Overall Study
Arm/Group | Iloprost
Started | 62
Completed | 11
Not Completed | 51
Not completed — Consent Withdrawal | 18
Not completed — Adverse Event | 7
Not completed — Serious Adverse Event | 13
Not completed — Non-compliance | 3
Not completed — Changed therapy | 2
Not completed — Patient received transplant | 2
Not completed — Patient had atrial septostomy | 1
Not completed — Patient weaned off iloprost | 1
Not completed — Mainly used Prodose not I-neb® device | 1
Not completed — Started intravenous prostacyclin | 1
Not completed — Started inhaled Remodulin | 1
Not completed — Patient had no improvement | 1

BASELINE CHARACTERISTICS:
Arm/Group | Iloprost
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 43
  >=65 years | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 52.5 (14.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Inhalation-times Rate - Iloprost PD-6 (Period I)
Description: Defined as the percentage of full doses (5 µg) of iloprost delivered within the recommended time frame for receiving a full dose of iloprost (4-10 minutes). Iloprost dosing information was available from the I-neb® device, which recorded the date and time of each inhalation, the duration of each inhalation, as well as the inhalation completion status (< 12.5%, ≥ 12.5% to < 100%, and Full)
Time Frame: 37 days prior to first dose of iloprost PD-15
Population: Modified intent-to-treat (MITT) population which includes all patients enrolled into the study who had at least 32 consecutive days of daily inhalation times data with PD-6, and at least 6 consecutive days of daily inhalation times data with PD-15.
Measure: Mean (Standard Deviation); unit: percentage of full doses administered
Groups:
- Iloprost PD-6: iloprost (10 µg/mL) standard dose (5 µg) delivered by I-neb® Adaptive Aerosol Delivery System (AAD) using Power Disc-6 (PD-6).
Arm/Group | Iloprost PD-6
Number analyzed (Participants) | 45
percentage of full doses administered | 29.9 (28.75)

2. Secondary Outcome: Number of Daily Inhalations - Iloprost PD-6 (Period I)
Description: Average number of daily inhalations. The number of daily inhalations was available from the I-neb® device, which recorded the date and time of each inhalation, the duration of each inhalation, as well as the inhalation completion status (< 12.5%, ≥ 12.5% to < 100%, and Full)
Time Frame: 37 days prior to first dose of iloprost PD-15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: inhalations/day
Arm/Group | Iloprost PD-6
Number analyzed (Participants) | 45
inhalations/day | 5.8 (1.22)

3. Secondary Outcome: Number of Daily Inhalations - Iloprost PD-15 (Period II)
Description: as for outcome 2
Time Frame: 37 days following first dose of iloprost PD-15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: inhalations/day
Groups:
- Iloprost PD-15: iloprost (10 µg/mL) standard dose (5 µg) delivered by I-neb® Adaptive Aerosol Delivery System (AAD) using Power Disc-15 (PD-15).
Arm/Group | Iloprost PD-15
Number analyzed (Participants) | 45
inhalations/day | 6.0 (1.11)

4. Secondary Outcome: Daily Inhalation Duration - Iloprost PD-6 (Period I)
Description: Average daily inhalation duration. The inhalation duration was available from the I-neb® device, which recorded the date and time of each inhalation, as well as the inhalation completion status (< 12.5%, ≥ 12.5% to < 100%, and Full)
Time Frame: 37 days prior to first dose of iloprost PD-15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Iloprost PD-6
Number analyzed (Participants) | 45
minutes | 15.0 (5.48)

5. Secondary Outcome: Daily Inhalation Duration - Iloprost PD-15 (Period II)
Description: as for outcome 4
Time Frame: 37 days following first dose of iloprost PD-15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Iloprost PD-15
Number analyzed (Participants) | 45
minutes | 7.2 (2.17)

6. Secondary Outcome: Percentage of Complete Doses Administered - Iloprost PD-6 (Period I)
Description: The frequency of dose completion was available from the I-neb® device, which recorded the date and time of each inhalation, the duration of each inhalation, as well as the inhalation completion status (< 12.5%, ≥ 12.5% to < 100%, and Full)
Time Frame: 37 days prior to first dose of iloprost PD-15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of complete doses
Arm/Group | Iloprost PD-6
Number analyzed (Participants) | 45
percentage of complete doses | 83.1 (21.18)

7. Secondary Outcome: Percentage of Complete Doses Administered - Iloprost PD-15 (Period II)
Description: as for outcome 6
Time Frame: 37 days following first dose of iloprost PD-15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of complete doses
Arm/Group | Iloprost PD-15
Number analyzed (Participants) | 45
percentage of complete doses | 98.0 (3.42)

8. Secondary Outcome: Percentage of Daily Doses Within the 6-9 Times/Day Treatment Regimen - Iloprost PD-6 (Period I)
Description: The frequency of daily inhalations was available from the I-neb® device, which recorded the date and time of each inhalation, the duration of each inhalation, as well as the inhalation completion status (< 12.5%, ≥ 12.5% to < 100%, and Full)
Time Frame: 37 days prior to first dose of iloprost PD-15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of daily doses
Arm/Group | Iloprost PD-6
Number analyzed (Participants) | 45
percentage of daily doses | 55.1 (29.53)

9. Primary Outcome: Inhalation-times Rate - Iloprost PD-15 (Period II)
Description: as for outcome 1
Time Frame: 37 days following first dose of iloprost PD-15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of full doses administered
Arm/Group | Iloprost PD-15
Number analyzed (Participants) | 45
percentage of full doses administered | 79.7 (17.45)

10. Secondary Outcome: Percentage of Daily Doses Within the 6-9 Times/Day Treatment Regimen - Iloprost PD-15 (Period II)
Description: as for outcome 8
Time Frame: 37 days following first dose of iloprost PD-15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of daily doses
Arm/Group | Iloprost PD-15
Number analyzed (Participants) | 45
percentage of daily doses | 66.1 (21.2)

11. Secondary Outcome: Systolic Blood Pressure - Iloprost PD-6 (Period I)
Description: SBP was recorded on Day 1 at 3 different timepoints: pre-inhalation, immediately post-inhalation and 15 minutes after inhalation of iloprost using PD-6
Time Frame: Day 1, prior to first dose of iloprost PD-15
Population: safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost PD-6
Number analyzed (Participants) | 62
mmHg
  pre-dose | 114.1 (11.68)
  immediately post-dose | 110.8 (11.47)
  15 minutes post dose | 113.0 (13.45)

12. Secondary Outcome: Systolic Blood Pressure (SBP) - Iloprost PD-15 (Day 1 and Day 7, Period II)
Description: SBP was recorded on Day 1 and Day 7 at 3 different timepoints: pre-inhalation, immediately post-inhalation and 15 minutes after inhalation of iloprost using PD-15
Time Frame: Day 1 and Day 7, following the first dose of iloprost PD-15
Population: safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost PD-15
Number analyzed (Participants) | 62
mmHg
  pre-dose (Day 1) | 114.5 (14.99)
  immediately post-dose (Day 1) | 111.7 (14.39)
  15 minutes post-dose (Day 1) | 113.9 (14.76)
  pre-dose (Day 7) | 114.7 (16.14)
  immediately post-dose (Day 7) | 109.7 (15.76)
  15 minutes post-dose (Day 7) | 113.1 (15.39)

13. Secondary Outcome: Diastolic Blood Pressure (DBP) - Iloprost PD-6 (Period I)
Description: DBP was recorded on Day 1 at 3 different timepoints: pre-inhalation, immediately post-inhalation and 15 minutes after inhalation of iloprost using PD-6
Time Frame: Day 1, prior to first dose of iloprost PD-15
Population: safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost PD-6
Number analyzed (Participants) | 62
mmHg
  pre-dose | 68.6 (10.94)
  immediately post-dose | 65.6 (8.98)
  15 minutes post-dose | 66.6 (9.79)

14. Secondary Outcome: Diastolic Blood Pressure (DBP) - Iloprost PD-15 (Day 1 and Day 7, Period II)
Description: DBP was recorded on Day 1 and Day 7 at 3 different timepoints: pre-inhalation, immediately post-inhalation and 15 minutes after inhalation of iloprost using PD-15
Time Frame: Day 1 and Day 7, following the first dose of iloprost PD-15
Population: safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Iloprost PD-15
Number analyzed (Participants) | 45
mmHg
  pre-dose (Day 1) | 67.5 (10.44)
  immediately post-dose (Day 1) | 65.2 (8.72)
  15 minutes post-dose (Day 1) | 67.9 (11.16)
  pre-dose (Day 7) | 68.6 (11.22)
  immediately post-dose (Day 7) | 65.7 (11.34)
  15 minutes post-dose (Day 7) | 66.7 (11.52)

15. Secondary Outcome: Heart Rate (HR) - Iloprost PD-6 (Period I)
Description: HR was recorded on Day 1 at 3 different timepoints: pre-inhalation, immediately post-inhalation and 15 minutes after inhalation of iloprost using PD-6
Time Frame: Day 1, prior to first dose of iloprost PD-15
Population: safety population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Iloprost PD-6
Number analyzed (Participants) | 62
beats per minute
  pre-dose | 79.2 (13.14)
  immediately post-dose | 78.9 (13.39)
  15 minutes post-dose | 76.1 (13.25)

16. Secondary Outcome: Heart Rate (HR) - Iloprost PD-15 (Day 1 and Day 7, Period II)
Description: HR was recorded on Day 1 and Day 7 at 3 different timepoints: pre-inhalation, immediately post-inhalation and 15 minutes after inhalation of iloprost using PD-15
Time Frame: Day 1 and Day 7, following the first dose of iloprost PD-15
Population: safety population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Iloprost PD-15
Number analyzed (Participants) | 62
beats per minute
  pre-dose (Day 1) | 78.0 (13.02)
  immediately post-dose (Day 1) | 77.9 (12.90)
  15 minutes post-dose (Day 1) | 76.4 (12.31)
  pre-dose (Day 7) | 77.8 (12.31)
  immediately post-dose (Day 7) | 78.3 (12.45)
  15 minutes post-dose (Day 7) | 76.0 (12.51)

17. Primary Outcome: Change in Inhalation-times Rate From Period I (Iloprost PD-6) to Period II (Iloprost PD-15)
Description: Change in the percentage of full doses (5 µg) of iloprost delivered within the recommended time frame for receiving a full dose of iloprost (4-10 minutes). Iloprost dosing information was available from the I-neb® device, which recorded the date and time of each inhalation, the duration of each inhalation, as well as the inhalation completion status (< 12.5%, ≥ 12.5% to < 100%, and Full)
Time Frame: 37 days prior to first dose of iloprost PD-15/37 days following first dose of iloprost PD-15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of full doses administered
Groups:
- Iloprost PD-15: iloprost (10 µg/mL) standard dose (5 µg) delivered by I-neb® Adaptive Aerosol Delivery System (AAD) using Power Disc-6 (PD-6) in Period I and Power Disc-15 (PD-15)in Period II.
Arm/Group | Iloprost PD-15
Number analyzed (Participants) | 45
percentage of full doses administered | 49.8 (34.28)
Statistical Analysis 1: Comparison: Iloprost PD-15; Comparison of the change in inhalation-times rate from Period I (PD-6) to Period II (PD-15); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = 49.8, 95% CI 2-sided [39.55 to 60.15]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline visit to end of study visit
Arm/Group | Iloprost PD-15
Serious Adverse Events (participants affected / at risk) | 27/62
Other Adverse Events (participants affected / at risk) | 53/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iloprost PD-15 (N=62)
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 10
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 3
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1
Right Ventricular Failure (Cardiac disorders) | 3
Cardiac Failure (Cardiac disorders) | 2
Acute Coronary Syndrome (Cardiac disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 1
Acute Right Ventricular Failure (Cardiac disorders) | 1
Atrial Tachycardia (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Coronary Artery Occlusion (Cardiac disorders) | 1
Bronchitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia Bacterial (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1
Reflux Oesophagitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 2
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 1
Fluid Overload (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Renal Failure (Renal and urinary disorders) | 2
Hepatitis (Hepatobiliary disorders) | 1
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 1
Liver Function Test Abnormal (Investigations) | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iloprost PD-15 (N=62)
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Headache (Nervous system disorders) | 7
Syncope (Nervous system disorders) | 6
Sinusitis (Infections and infestations) | 8
Upper Respiratory Tract Infection (Infections and infestations) | 7
Urinary Tract Infection (Infections and infestations) | 5
Nausea (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 13
Chest Pain (General disorders) | 7
Oedema (General disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 9
Fluid Retention (Metabolism and nutrition disorders) | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Palpitations (Cardiac disorders) | 6
International Normalised Ratio Increased (Investigations) | 5
Flushing (Vascular disorders) | 5
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4

LIMITATIONS AND CAVEATS:
Study was terminated early due to the discontinuation of the I-neb Power Disc-15 development program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No